CLINICAL TRIAL: NCT05574075
Title: Assessment of Motor Adaptation in Precision Grip Performance of Children: a Kinetic Analysis of Responsive Grip Behavior
Brief Title: Assessment of Motor Adaptation in Precision Grip Performance of Children
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B-BR-110-072
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Hand Strength, Child, Sensation, White Matter
Keywords: Hand Strength, Child, Sensation, White matter
MeSH Terms: interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- group of preterm and term children: group 1: preterm children group 2: term children
  Interventions: Diagnostic Test: Diffusion tensor imaging
- group of different ages of preschool children: group 1: children with age of 25 months-36 months group 2: children with age of 37 months-48 months group 3: children with age of 49 months-60 months

INTERVENTIONS:
Diagnostic Test: Diffusion tensor imaging — white matter imaging markers
  Groups: group of preterm and term children

SUMMARY:
Preterm children usually suffer from mild hand motor performance, however, the problem are rarely detected in time. Identifying the pathology causing deficits in sensorimotor control of a hand helps the occupational therapist to determine appropriate clinical decision-making for intervention. Well-motor performance requires complete sensorimotor control. Understanding hand sensorimotor control mechanism and its neural control can help clinicians find the reason behind hand motor deficits. The analysis of motion adaptation of the precision pinch behavior in the perturbing environment has been regarded as a clinically meaningful tool for evaluating sensorimotor control of a hand, especially for the complex anatomical structure of bone and tendon. The motor adaptation analysis for the precision grip behavior can provide the temporal and spatial parameters of dynamic grip force adjustment. Therefore, the exploration of motor adjustment can provide in-depth understanding of the neural mechanisms that lead to impairment of motor function and skill acquisition of a child, which can assist clinical occupational therapist in identifying the cause and severity of impairment of children's hand skills and provide appropriate strategies and types of treatment. The recent research on children's motor adaptation focuses on the discussion of the efficiency of motor adaptation in unfamiliar or disturbing task situations. Thus, the first purpose of this research is to develop an easy-to-detect apparatus to detect the adjustment efficiency of a responsive grip behavior of children in a disturbing pinch-lifting task and to construct the reliability of its evaluation. The second purpose of the research is to understand the correlation between the efficiency of children's reactive pinch performance adjustment and the results of traditional evaluation of fine motor development scale and sensorimotor control assessments. The third purpose of the research is to analyze the difference in motor adjustment of a precision pinch performance at different ages of preschool children. The fourth purpose is to compare the efficiency of motor adaptation in preterm and term children. In addition, preterm birth is often accompanied by white matter abnormalities and affects future hand motor performance. Investigating white matter imaging markers for predicting motor adaptation can help early detection of problems. Therefore, the fifth objective was to explore whether specific white matter imaging markers can predict the efficiency of reactive motor adaptation.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to do reach-to-grasp performance
2. Intact comprehension ability

Exclusion Criteria:

1. Diagnosis of cerebral palsy and other genetic or congenital damage
2. Bone and nerve damage in the upper limbs in the past year
3. Un-correctable problems of vision or hearing impairment

Ages: 2 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: healthy adults: 20-39 years old term children: 24-60 months preterm children: 24-48 months
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
responsive grip behavior | up to 2 years
  amplitude of pinch force development or adaptation to perturbation

SECONDARY OUTCOMES:
The Bayley Scales of Infant and Toddler Development, Third Edition | up to 2 years
  for diagnosing developmental delays in early childhood
Peabody Developmental Motor Scales, Second Edition | up to 2 years
  measure interrelated motor abilities of children from birth through age 5 years of age
Tuning Fork 128 Hz | up to 2 years
  measure vibration sense
Box and blocks test | up to 2 years
  measure upper limb coordination
Semmes-Weinstein monofilament test | up to 2 years
  measure touch-pressure sense

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsu HY, Yu JN, Lin YC, Su HC, Koh CL, Kuo LC. Impact of hemispheric specialization on reactive upper limb motor control after perturbations via a newly designed reactive pinch-holding-up activity test. Clin Biomech (Bristol). 2025 Aug;128:106607. doi: 10.1016/j.clinbiomech.2025.106607. Epub 2025 Jul 4. PMID 40633224